CLINICAL TRIAL: NCT06006936
Title: Testing the Efficacy of the 'Coping With Infertility' Self-Help Program: A Randomized Controlled Trial
Brief Title: Testing an Evidence-Based Self-Help Program for Infertility-Related Distress in Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Regina (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Saskatchewan Health Research Foundation (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Jennifer Gordon, Associate Professor, University of Regina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB #2023-210; DCO150GP (Other Grant/Funding Number: Canadian Institutes of Health Research); 6447 (Other Grant/Funding Number: Saskatchewan Health Research Foundation)
Record Dates: First submitted 2023-08-17; First posted 2023-08-23 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Infertility; Distress, Emotional; Mental Health Issue
Keywords: infertility; women; mental health; distress; quality of life; depression; anxiety; relationship quality; randomized controlled trial; intervention; treatment; self-help
MeSH Terms: conditions — Infertility; Psychological Well-Being; Depression; Anxiety Disorders | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either receive the CWI program or to remain in a treatment-as-usual (TAU) control condition using stratified block randomization. The two arms will be stratified based on whether participants are attempting to conceive naturally or undergoing fertility treatments.
  Participants in the intervention condition will receive one 10-minute video module from the CWI program every week for seven weeks. Each video module will include a homework assignment encouraging participants to integrate the module content into everyday life.
  Participants in the TAU control condition will not receive video modules or homework; instead, they will continue with everyday life-including their attempts to conceive-until the conclusion of the study. TAU participants will be offered the intervention following the conclusion of the study.
Who Masked: Outcomes Assessor
Masking Description: A research assistant (RA) who is not involved with this study will use the randomization scheme to prepare opaque envelopes with each participant's treatment assignment, to be opened at the end of each enrolment session. While it is not possible to maintain full blinding of either the participant or the researchers given the nature of the intervention, all outcomes will be collected by an RA who is blind to participants' treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Condition (Experimental): This arm will receive the Coping with Infertility intervention.
  Interventions: Behavioral: Coping with Infertility Self-Help Program
- Waitlist/Treatment as Usual Control Condition (No Intervention): This arm will continue with everyday life-including their attempts to conceive.

INTERVENTIONS:
Behavioral: Coping with Infertility Self-Help Program — The CWI program consists of seven 10-minute videos, each with accompanying homework assignments.
  The first module, cognitive restructuring, includes instructions on challenging extreme or unhelpful automatic thoughts. The second module, challenging negative core beliefs, includes looking for patterns in thinking that illustrate core beliefs. The third module features behavioural activation techniques and emphasizes the importance of regular pleasure and skill-based activities. The fourth module highlights coping with grief and factors that contribute to grief, such as individual differences in grieving style. The fifth module supports strengthening relationships through responding to requests for affection and outlines several common relationship mistakes. The sixth module demonstrates how to identify and use values to make decisions and guide behaviour. The seventh module summarizes how thoughts, actions, and interactions can contribute to well-being when experiencing infertility.
  Arms: Intervention Condition

SUMMARY:
Now affecting one in six couples in Canada, infertility is defined as a lack of conception after 12 or more months of regular, unprotected sexual intercourse. Infertility can result from a number of causes; however, women are responsible for accommodating rigid treatment regimens and carry a disproportionate share of the psychological burden associated with infertility. Thirty to forty percent of women presenting for the evaluation of infertility experiencing clinically significant depression or anxiety. Yet access to infertility-specific mental health resources is extremely limited in Canada; current psychological interventions are not specialized to this population and are largely ineffective at reducing distress. Therefore, there is an enormous need to increase the efficacy and accessibility of mental health resources for this population.

To address this need, the 7-week Coping with Infertility (CWI) program was developed in collaboration with women with lived experience with infertility. The CWI program aims to reduce distress related to infertility and was recently tested in a small pilot study, where it was found to be very effective in reducing depression and anxiety and improving quality of life among individuals struggling to get pregnant. The goal of this clinical study is to test the CWI program in adult women experiencing infertility. The main questions it aims to answer are if the CWI program is effective at improving mental health and well-being in women experiencing infertility, and if demographic or lifestyle factors moderate the effect of the treatment. For seven weeks, participants will receive the CWI program and complete online questionnaires and interviews to assess the program's effects on infertility-related distress, quality of life, depressive symptoms, anxiety, and relationship quality. They will then complete these questionnaires biweekly for 16 weeks following the program. Researchers will compare the CWI program to a waitlist/treatment as usual control condition to see if the program reduces psychological distress above and beyond women's ordinary coping strategies. If the program is effective in improving psychological well-being in this clinical study, the researchers will make the program widely and freely available to women throughout Canada and the world.

DETAILED DESCRIPTION:
Infertility is associated with severe psychological consequences; psychiatric disorders are common, particularly in women, yet current psychological interventions are not specialized to this population and are largely ineffective. The 7-week Coping with Infertility (CWI) program is a self-help program based on cognitive behaviour therapy that aims to improve mental health in women and individuals assigned female at birth who are experiencing infertility. This study aims to test the efficacy of the CWI program.

In the proposed study, a single-blind randomized controlled trial, participants will be randomly assigned to either the specialized CWI program or a waitlist/treatment as usual control condition using stratified block randomization. Infertility-related distress, quality of life, depression, anxiety, and relationship quality will be assessed at baseline, midway through the program, post-treatment, and biweekly for 16 weeks after treatment. It is expected that participants assigned to the CWI program will show significantly reduced infertility-related distress, depression, and anxiety, and improved quality of life and relationship quality relative to baseline and the waitlist control condition. Moderation analyses will examine potential treatment moderators including sexual orientation and gender identity, as well as cultural background, disability status, and whether participants are pursuing fertility treatments. Participants who complete the CWI program will also provide qualitative feedback on how the program can be improved. The results of this trial could establish the CWI program as an effective short-term therapy option for women experiencing infertility, addressing a significant gap in infertility treatment.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* Experiencing infertility (defined as [a] lack of conception after 12 or more months of regular, unprotected, heterosexual intercourse, or [b] currently undergoing fertility treatments)
* Fluent in English

Exclusion Criteria:

* Under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fertility Quality of Life (FertiQoL) Score, at Mid-Treatment, Post-Treatment and Biweekly for 16 Weeks Post-Treatment | 6 months (FertiQoL completed midway through the program (week 4), post-program (week 8), then biweekly up to 16 weeks after the end of treatment)
  Fertility-related quality of life will be measured via the 24 items contained within the core FertiQoL scale. Scores range from 0 to 100; participants will be considered to exhibit significantly poorer quality of life if their FertiQoL score is less than or equal to 71.

SECONDARY OUTCOMES:
Mean Infertility-Related Distress Scores on the Copenhagen Multi-Centre Psychosocial Infertility - Fertility Problem Stress Scales (COMPI-FPSS), at Post-Treatment and Biweekly for 16 Weeks Post-Treatment | 6 months (COMPI-FPSS completed midway through the program (week 4), post-program (week 8), then biweekly up to 16 weeks after the end of treatment)
  Infertility-related distress will be measured via the nine items contained within the COMPI-FPSS. Scores range from 9 to 38; higher scores indicate greater distress.
Mean Depression Scores on the Patient Health Questionnaire-9 (PHQ-9), at Post-Treatment and Biweekly for 16 Weeks Post-Treatment | 6 months (PHQ-9 completed midway through the program (week 4), post-program (week 8), then biweekly up to 16 weeks after the end of treatment)
  Depressive symptoms will be measured via the nine items contained within the PHQ-9. Scores range from 0 to 27; participants will be considered to exhibit major depressive disorder if their PHQ-9 score is greater than or equal to 10.
Mean Anxiety Scores on the Generalized Anxiety Disorder-7 (GAD-7), at Post-Treatment and Biweekly for 16 Weeks Post-Treatment | 6 months (GAD-7 completed completed midway through the program (week 4), post-program (week 8), then biweekly up to 16 weeks after the end of treatment)
  Anxious symptoms will be measured via the seven items contained within the GAD-7. Scores range from 0 to 21; participants will be considered to exhibit generalized anxiety disorder if their GAD-7 score is greater than or equal to 10.
Mean Relationship Quality on the Relationship Assessment Scale (RAS), at Post-Treatment and Biweekly for 16 Weeks Post-Treatment | 6 months (RAS completed midway through the program (week 4), post-program (week 8), then biweekly up to 16 weeks after the end of treatment)
  Relationship quality will be measured via the seven items contained within the RAS. Scores range from 7 to 35; higher scores indicate greater relationship stability, satisfaction, and quality while lower scores indicate greater relationship dissatisfaction and distress. Participants will be considered to exhibit relationship dissatisfaction and distress if their average RAS score is less than four.
Occurrence of Mood and Anxiety Disorders at Baseline, Post-Treatment, and 16 Weeks After Treatment | 6 months (NetSCID completed at enrollment (week 0), post-program (week 8), and 16 weeks after the end of treatment)
  The presence or absence of major depressive disorder, persistent depressive disorder, generalized anxiety disorder, and panic disorder will be determined using the Computerized Version of the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (NetSCID). Presence of any mood and anxiety disorders will be simultaneously and automatically calculated by the NetSCID system based on the relevant criteria results.

OTHER OUTCOMES:
Mean Intervention Credibility and Participant Expectancy at Baseline, Using the Credibility and Expectancy Questionnaire (CEQ) | CEQ completed at enrollment (week 0)
  Intervention credibility and participant expectancy will be measured via the six items contained within the CEQ. Scores range from 3 to 27 for each of the two subscales; higher scores indicate greater program credibility and participant expectancy.
Mean Quality of Homework Completion on the Homework Rating Scale (HRS) | 7 weeks (HRS completed weekly throughout the program)
  Homework compliance will be measured via the 12 items contained within the HRS. Scores range from 0 to 36; higher scores indicate better quality and quantity of completion.
Mean Treatment Acceptability Post-Treatment, Using the Treatment Acceptability/Adherence Scale (TAAS) | TAAS completed one week after the end of treatment (week 8)
  Intervention acceptability will be measured via the 10 items contained within the TAAS. Scores range from 10 to 70; higher scores indicate greater program acceptability and adherence.
Mean Adverse Events Perceived to be Related to the Intervention Post-Treatment, Using the Negative Effects Questionnaire (NEQ) | NEQ completed one week after the end of treatment (week 8)
  Potential adverse events perceived to be related to the intervention will be measured via the 20 items contained within the NEQ. Items will be summed to determine the number of negative effects participants have experienced, divided by whether they believe the experience was caused by the treatment or other circumstances; higher scores indicate more negative effects attributed to the intervention.
Mean Healthcare Utilization, Medical and Productivity Costs in the 16 Weeks After Treatment, Using the Treatment Inventory of Costs in Patients with Psychiatric Disorders (TiC-P) | TiC-P completed 16 weeks after the end of treatment (week 24)
  Participants' healthcare utilization will be measured via the 33 items contained within the TiC-P. An additional section has been added to specifically ask about receipt of fertility treatments. Direct medical costs incurred by participants during the 16 weeks post-treatment will be calculated by multiplying the number of appointments participants have had with different general healthcare and mental healthcare professionals by the unit cost of these services in Canada. Similarly, productivity costs incurred during the 16 weeks post-treatment will be calculated by multiplying the number of hours of productivity lost to absenteeism or reduced efficiency by a standard cost price of productivity (e.g., $30 CAD per hour).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L. Gordon, Ph.D., Principal Investigator — Unviersity of Regina
Locations (1):
- University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Poulter MML, Wahl TD, Kiviharju MJ, Campbell TS, Gordon JL. Testing the efficacy of a self-guided psychotherapy intervention for infertility-related distress: a randomized controlled trial. Hum Reprod. 2025 Dec 16:deaf237. doi: 10.1093/humrep/deaf237. Online ahead of print. PMID 41401817
- [Derived] Gordon JL, Poulter MML, Balsom AA, Campbell TS. Testing an Evidence-Based Self-Help Program for Infertility-Related Distress: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Jan 18;13:e52662. doi: 10.2196/52662. PMID 38236638